CLINICAL TRIAL: NCT05664230
Title: Efficacy of Osteopathic Treatment on the Side Effects of Curative Treatments of Lymphoblastic Leukemia in Pediatrics
Acronym: Leucosteo
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP220699; IDRCB: 2022-A01261-42 (Registry Identifier: French Health Authority)
Record Dates: First submitted 2022-12-07; First posted 2022-12-23 (Actual); Last update posted 2022-12-23 (Actual); Status verified 2022-10

CONDITIONS: Lymphoblastic Leukemia
Keywords: osteopathy
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Osteopathic Physicians

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: osteopathy — five osteopathy sessions
  Other Names: osteopathy session

SUMMARY:
During the curative treatment of cancer, pain often remains the dominant symptom affecting the physical and psychological state of the patient.

Osteopathy is an exclusively manual practice whose goal is to compensate for mobility dysfunctions of the tissues of the human body. It can be used as a complementary treatment for cancer pain when pain medications are not enough.

The aim of this study is to examine the effectiveness of osteopathy in reducing pain intensity and improving quality of life in patients treated for pediatric acute lymphoblastic leukemia.

DETAILED DESCRIPTION:
During the curative treatment of cancer, pain often remains the dominant symptom affecting the physical and psychological state of the patient.

Osteopathy is an exclusively manual practice whose goal is to compensate for mobility dysfunctions of the tissues of the human body. It can be used as a complementary treatment for cancer pain when pain medications are not enough.

The aim of this study is to examine the effectiveness of osteopathy in reducing pain intensity and improving quality of life in patients treated for pediatric acute lymphoblastic leukemia.

Primary objective :

To evaluate the effectiveness of five osteopathy sessions at regular intervals on the characteristics of the pain felt in patients aged 1 to 10 years treated for acute lymphoblastic leukemia using the HEDEN scale (Hetero-Evaluation Pain Child).

ELIGIBILITY:
Inclusion Criteria:

* Patient managed and treated with a diagnosis of acute lymphoblastic leukemia
* Patient between 1 and 10 years of age
* Patient with pain at inclusion, or pain at diagnosis related to leukemia
* Social security affiliation or entitlement
* Signature of informed consent by both parents

Exclusion Criteria:

* No pain reported at the time of management or diagnosis
* Surgery less than 30 days old
* Patient with another contraindication to osteopathic treatment (worsening of the condition, bleeding syndrome), or a psychiatric pathology that prevents the scales from being used.

Ages: 1 Year to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients with acute lymphoblastic leukemia
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2023-01-01 (Estimated); Primary Completion 2023-07-01 (Estimated); Study Completion 2023-08-01 (Estimated)

PRIMARY OUTCOMES:
Evaluate the effectiveness of 5 weekly osteopathy sessions at regular intervals from week 1 to week 5 on the characteristics of the pain felt in patients aged 1 to 10 years treated for acute lymphoblastic leukemia using the HEDEN scale. | 5 weeks
  HEDEN (Hetero-Evaluation Pain Child) score before and after each intervention

SECONDARY OUTCOMES:
Evaluate the effectiveness of 5 weekly osteopathy sessions at regular intervals from week 1 to week 5 on the intensity of the pain felt in patients aged 4 to 10 years treated for acute lymphoblastic leukemia using the face scale: FPS -R. | 5 weeks
  FPS-R (Face Pain Scale-Revised) score before and after each osteopathy session
To study the variations in quality of life at inclusion and at the end of the study using the PedsQL™ (questionnaire quality of life in paediatrics). | 5 weeks
  PedsQL™ Questionnaire quality of life in paediatrics

CONTACTS AND LOCATIONS:
Overall Officials: Benoit BRETHON, MD, Principal Investigator — Assistant Publique Hopitaux de Paris
Locations (1):
- Robert Debré Hospital, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided